CLINICAL TRIAL: NCT04525807
Title: Precision Medicine for Colorectal Cancer Liver Metastasis Guided by Multi-omics Data Under the Umbrella Theory
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-08
Record Dates: First submitted 2020-08-21; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiomics arm: Guide therapy based on multi-omics
  Interventions: Diagnostic Test: Multi-omics

INTERVENTIONS:
Diagnostic Test: Multi-omics — Use multi-omics to analyze

SUMMARY:
In order to more accurately discover the cause of drug resistance in tumor treatment, and to provide a new basis for precise treatment.

Therefore, based on the umbrella theory of precision medicine, we carried out this single-center, prospective, and observational study to include patients with liver metastases from colorectal cancer. By combining genome, transcriptome, and proteomic sequencing data, we established a basis for colorectal cancer liver Transfer the multi-omics data of the sample, describe the reason for the resistance of the first-line treatment, and search for new therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* ECOG score 0-2 points
* Pathologically diagnosed patients with colorectal cancer
* Combined with liver metastases confirmed by imaging, and the lesion is measurable (RECIST standard)
* The lesion is available
* First-line treatment failed; hematology, liver and kidney function tests are suitable for back-line treatment
* Informed consent

Exclusion Criteria:

* With brain metastases
* History of other malignancies
* Pregnancy or breastfeeding
* Have received other drug clinical studies within 30 days before the start of this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were newly diagnosed with liver metastases from colorectal cancer (pathologically diagnosed as adenocarcinoma)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 1 year
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including complete remission (CR) and partial remission (PR) cases

SECONDARY OUTCOMES:
progression-free survival | 1 year
  Refers to the date from initial diagnosis to tumor progression
Overall survival | 3 years
  Refers to the date from initial diagnosis to last follow-up or death date

IPD SHARING:
Plan to Share IPD: No